CLINICAL TRIAL: NCT06891573
Title: A Multicenter, Feasibility Randomized Controlled Study to Evaluate the Applicability and Safety of the Software 'SUPERAGING' for Cognitive Therapy and Musculoskeletal Analysis in Frail or Prefrail Patients
Brief Title: South Korean Study to Prevent Frailty and Aging-related Diseases Through Lifestyle Intervention
Acronym: SUPERAGING
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Seong Hye Choi, MD (Other)
Responsible Party: Sponsor-Investigator, Seong Hye Choi, MD, Professor, Inha University Hospital
Organization: Inha University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024-07-020
Record Dates: First submitted 2025-02-25; First posted 2025-03-24 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Frailty
Keywords: frailty; intervention; multidomain; digital
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Participants will receive interventions including exercise, cognitive training, nutrition education, and management of diseases related to frailty via the app for one hour per day, five days a week for 16 weeks.
  Interventions: Behavioral: Lifestyle Management
- Control (No Intervention): Participants in the control group will receive standard treatment related to frailty during the study period and be provided with guidelines on 'Lifestyle habits for treating frailty or prefrailty'.

INTERVENTIONS:
Behavioral: Lifestyle Management — For 16 weeks, participants will receive exercise, cognitive training, nutrition education, and disease education through a smartphone app, and the content and intensity of the intervention will be adjusted every four weeks through an assessment of frailty symptoms through the app.
  Arms: Intervention group

SUMMARY:
The goal of this feasibility randomized controlled trial is to investigate the applicability of software that aims to improve symptoms of frailty by implementing customized interventions such as physical exercise and cognitive training implemented through a mobile app for 16 weeks for patients diagnosed with frailty or prefrailty. The primary outcomes are adherence, retention rates, and recruitment rates. Participants will participate in customized interventions including physical exercise, cognitive training, nutritional guidance, and management of disease related to frailty for 16 weeks.

DETAILED DESCRIPTION:
The physical exercise program will comprise aerobic exercise, balance-improving exercises, flexibility-enhancing activities, and strength-building exercises targeting major muscle groups through a mobile app . Customized cognitive training, performed using a mobile app, targets the cognitive domains of prospective memory and executive function. Nutritional intervention will be performed to treat frailty symptoms and disease related to frailty through a mobile app. Education and management of disease related to frailty will be done through a mobile app.

ELIGIBILITY:
Inclusion Criteria:

* 60-90 years of age
* Residing in the community
* Total score of Modified Fried frailty phenotype score ≥ 1 point
* Korean Mini-Mental State Examination-2 z-score ≥ -1.5
* Can read and write
* Being able to use the a mobile app through education or having someone help a participant use the mobile app
* Having a reliable informant who could provide investigators with the requested information.
* written informed consent

Exclusion Criteria:

* Major psychiatric illness such as major depressive disorders
* Dementia
* Other neurodegenerative disease (e.g., Parkinson's disease)
* Malignancy within five years
* Cardiac stent or revascularization within one year
* Serious or unstable symptomatic cardiovascular disease
* Other serious or unstable medical disease such as acute or severe asthma, active gastric ulcer, severe liver disease, or severe renal disease
* Severe loss of vision, hearing, or communicative disability
* Significant laboratory abnormality that may result in cognitive impairment
* Any conditions preventing cooperation as judged by the study physician
* Unable to participate in exercise program safely
* Coincident participation in any other intervention trial

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-02-26 (Actual); Primary Completion 2025-12-20 (Estimated); Study Completion 2026-01-15 (Estimated)

PRIMARY OUTCOMES:
retention rate | From enrollment to the end of intervention at 16 weeks
  retention rate ≥ 70%
Adherence to the protocol | From enrollment to the end of intervention at 16 weeks
  Adherence to the protocol ≥ 70%
recruitment rate | From enrollment to the end of intervention at 16 weeks
  recruitment rate ≥ 50%.

SECONDARY OUTCOMES:
Change from Baseline in Korean Frailty Index for Primary Care at 16 weeks | From baseline to the end of intervention at 16 weeks
  The score ranges from 0 to 1. A lower score indicates better performance.
Change from Baseline in Modified Fried frailty phenotype score at 16 weeks | From baseline to the end of intervention at 16 weeks
  The score ranges from 0 to 5. A lower score indicates better performance.
Change from Baseline in Lubben Social Network Scale at 16 weeks | From baseline to the end of intervention at 16 weeks
  The score ranges from 0 to 50. A higher score indicates better performance.
Change from Baseline in 14-item cognitive subscale of the Alzheimer's Disease Assessment Scale at 16 weeks | From baseline to the end of intervention at 16 weeks
  The score ranges from 0 to 90. A lower score indicates better performance.
Change from Baseline in Korean Mini-Mental State Examination-2 at 16 weeks | From enrollment to the end of intervention at 16 weeks
  The score ranges from 0 to 30. A higher score indicates better performance.
Change from Baseline in Clinical Dementia Rating scale-Sum of Boxes at 16 weeks | From baseline to the end of intervention at 16 weeks
  The score ranges from 0 to 18. A lower score indicates better performance.
Change from Baseline in Korean Instrumental Activities of Daily Living at 16 weeks | From baseline to the end of intervention at 16 weeks
  The score ranges from 0 to 3. A lower score indicates better performance.
Change from Baseline in Modified Barthel Index: at 16 weeks | From baseline to the end of intervention at 16 weeks
  The score ranges from 0 to 100. A higher score indicates better performance.
Change from Baseline in Center for Epidemiological Studies-Depression Scale at 16 weeks | From baseline to the end of intervention at 16 weeks
  The score ranges from 0 to 60. A lower score indicates better performance.
Change from Baseline in Quality of life-Alzheimer's disease at 16 weeks | From baseline to the end of intervention at 16 weeks
  The score ranges from 0 to 52. A higher score indicates better performance.
Change from Baseline in gait speed at 16 weeks | From baseline to the end of intervention at 16 weeks
  A lower score indicates better performance.
Change from Baseline in Short Physical Performance Battery at 16 weeks | From baseline to the end of intervention at 16 weeks
  The score ranges from 0 to 12. A higher score indicates better performance.
Change from Baseline inTimed Up and Go test at 16 weeks | From baseline to the end of intervention at 16 weeks
  A lower score indicates better performance.
Change from Baseline in 30 s sit-to-stand at 16 weeks | From baseline to the end of intervention at 16 weeks
  A higher score indicates better performance.
Change from Baseline in 2 min stepping test at 16 weeks | From baseline to the end of intervention at 16 weeks
  A higher score indicates better performance.
Change from Baseline in Mini Nutritional Assessment at 16 weeks | From baseline to the end of intervention at 16 weeks
  The score ranges from 0 to 14. A higher score indicates better performance.
Change from Baseline in Nutritional Quotient for Elderly at 16 weeks | From baseline to the end of intervention at 16 weeks
  The score ranges from 0 to 100. A higher score indicates better performance.
Change from Baseline in skeletal muscle mass at 16 weeks | From baseline to the end of intervention at 16 weeks
  A higher score indicates better performance.
Number of Participants with Treatment-Related Adverse Events | From enrollment to the end of intervention at 16 weeks
  A lower score indicates better performance.
Change from baseline in MIND diet checklist at 16 weeks | From baseline to the end of intervention at 16 weeks
  The score ranges from 0 to 15. A higher score indicates better performance.
Change from baseline in International Physical Activity Questionnaire-Short Form at 16 weeks | From baseline to the end of intervention at 16 weeks
  The score ranges from 0 to 20,000. A higher score indicates better performance.
Change from baseline in LDL-C at 16 weeks | From baseline to the end of intervention at 16 weeks
  The score ranges from 0 to 300. A lower score indicates better performance.
Change from baseline in HDL-C at 16 weeks | From baseline to the end of intervention at 16 weeks
  The score ranges from 0 to 200. A higher score indicates better performance.
Change from baseline in HbA1c at 16 weeks | From baseline to the end of intervention at 16 weeks
  The score ranges from 0 to 30. A lower score indicates better performance.
Change from baseline in eGFR at 16 weeks | From baseline to the end of intervention at 16 weeks
  The score ranges from 0 to 200. A higher score indicates better performance.
Change from baseline in blood pressure at 16 weeks | From baseline to the end of intervention at 16 weeks
  The score ranges from 0 to 250. A lower score indicates better performance.
Change from baseline in body weight at 16 weeks | From baseline to the end of intervention at 16 weeks
  The score ranges from 0 to 200. A higher score indicates better performance in frailty.
Change from baseline in waist circumference at 16 weeks | From baseline to the end of intervention at 16 weeks
  The score ranges from 0 to 200. A higher score indicates better performance in frailty.
Occurrence of aging-related diseases | From baseline to the end of intervention at 16 weeks
  The score ranges from 0 to 10. A lower score indicates better performance.

CONTACTS AND LOCATIONS:
Overall Officials: Seong Hye Choi, MD, PhD, Principal Investigator — Inha University Hospital
Locations (3):
- South Korea (3):
  - Inha University Hospital, Incheon
  - Ewha Womans University Seoul hospital, Seoul
  - Ajou University Hospital, Suwon

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data will be shared with the Global Alzheimer's Association Interactive Network.
Supporting Information: Study Protocol, SAP
Time Frame: The data will become in 2027 and become available for 5 years.
Access Criteria: The access criteria is an approval of steering committee.

REFERENCES:
- [Derived] Jung S, Kang HJ, Moon SY, Choi M, Jung J, Kim HR, Jung S, Jeong JH, Choi SH, Park YK. South Korean study to prevent the progression of frailty and aging-related diseases using a digital multidomain intervention (SUPERAGING): Protocol of a feasibility pilot study. Digit Health. 2026 Jan 6;12:20552076251410995. doi: 10.1177/20552076251410995. eCollection 2026 Jan-Dec. PMID 41509872